CLINICAL TRIAL: NCT01163149
Title: A Randomized, Open-Label, Multicenter, Multinational, Dose-Ranging, Concurrent Control Study of the Safety, Efficacy, Pharmacokinetic of ENB-0040 (Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein) in Adolescents and Adults With Hypophosphatasia (HPP)
Brief Title: Safety and Efficacy Study of Asfotase Alfa in Adolescents and Adults With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENB-009-10
Record Dates: First submitted 2010-06-24; First posted 2010-07-15 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; Bone Disease; Soft Bones; Low Alkaline Phosphatase; genetic metabolic disorder; alkaline phosphatase; tissue-specific alkaline phosphatase (TNSALP); rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Cohort 1: Daily SC injections of 0.3 mg/kg asfotase alfa (2.1 mg/kg/week total)
  Interventions: Drug: asfotase alfa
- Cohort 2 (Experimental): Cohort 2: Daily SC injections of 0.5 mg/kg asfotase alfa (3.5 mg/kg/week total)
  Interventions: Drug: asfotase alfa
- Concurrent Control (No Intervention): Following completion of the Week 24 visit, all patients (including those randomized to the concurrent control cohort) may be eligible to participate in an open-label extension treatment period. In this extension period, all patients will be treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects will receive 1 mg/kg/day 6 days/week for an additional 48 weeks or until regulatory approval of the drug.

INTERVENTIONS:
Drug: asfotase alfa — Cohort 1: Daily SC injections of 0.3 mg/kg asfotase alfa (total of 2.1 mg/kg/week)
  Arms: Cohort 1
Drug: asfotase alfa — Cohort 2: Daily SC injections of 0.5 mg/kg Asfotase Alfa (3.5 mg/kg/week total)
  Arms: Cohort 2

SUMMARY:
This clinical trial was conducted to study hypophosphatasia (HPP), a bone disorder caused by gene mutations or changes. These gene mutations cause low levels of an enzyme needed to harden bone. The purpose of this study was to test the safety and efficacy of two doses of the study drug called asfotase alfa as compared to a control group to see effects on adolescents and adults with HPP.

DETAILED DESCRIPTION:
Asfotase alfa was formerly referred to as ENB-0040

Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

* Patients or their legal representative(s) must provide written informed consent prior to undergoing any study-related procedures
* Patients must be ≥ 13 and ≤ 65 years of age at the time of study enrollment
* Female patients of childbearing potential and sexually mature males must agree to use a medically acceptable form of birth control; for the purposes of this study, females are considered of non-childbearing potential if they are surgically sterile (i.e., have undergone a total hysterectomy, bilateral salpingo-oophorectomy or tubal ligation) or are post-menopausal, defined as having complete cessation of menstruation for at least 1 year after 45 years of age
* Patients must have a pre-established clinical diagnosis of HPP as indicated by:

  * Serum alkaline phosphatase (ALP) below the age-adjusted normal range
  * Plasma PLP at least twice the upper limit of normal (no vitamin B6 administered for at least 1 week prior to determination)
  * Evidence of osteopenia or osteomalacia on skeletal radiographs
* Patients must have osteomalacia on bone biopsy, characterized by an MLT z-score of +2 or more (results from ENB-001-08 may be used)
* Patients must be willing to comply with study procedures and the visit schedule

Exclusion criteria:

Patients will be excluded from participation in this study if they meet any of the following exclusion criteria:

* Women who are pregnant or lactating
* History of sensitivity to tetracycline
* Serum calcium or phosphate levels below the normal range
* Serum 25(OH) vitamin D below 20 ng/mL
* Serum creatinine or parathyroid hormone (PTH) levels above the upper limit of normal
* Medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities
* Orthopedic surgery within 12 months prior to study entry that may interfere with the ability to perform functional assessments for the study
* Prior treatment with bisphosphonates within 2 years of study entry for any length of time or for more than 2 years at any time point; for patients with prior bisphosphonate use that is allowed, the bone resorption markers serum C-telopeptide and urine N-telopeptide or urine deoxypyridinoline must also be within the normal range or elevated to be eligible for study participation
* Treatment with PTH within 6 months prior to the start of asfotase alfa administration
* Participation in an interventional or investigational drug study within 30 days prior to study participation

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Shriner's Hospital for Children, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
- Health Sciences Centre Winnipeg, University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Millan JL, Narisawa S, Lemire I, Loisel TP, Boileau G, Leonard P, Gramatikova S, Terkeltaub R, Camacho NP, McKee MD, Crine P, Whyte MP. Enzyme replacement therapy for murine hypophosphatasia. J Bone Miner Res. 2008 Jun;23(6):777-87. doi: 10.1359/jbmr.071213. PMID 18086009
- [Derived] Simmons JH, Rush ET, Petryk A, Zhou S, Martos-Moreno GA. Dual X-ray absorptiometry has limited utility in detecting bone pathology in children with hypophosphatasia: A pooled post hoc analysis of asfotase alfa clinical trial data. Bone. 2020 Aug;137:115413. doi: 10.1016/j.bone.2020.115413. Epub 2020 May 14. PMID 32417537
- [Derived] Gospe SM 3rd, Santiago-Turla C, DeArmey SM, Cummings TJ, Kishnani PS, Bhatti MT. Ectopic Ocular Surface Calcification in Patients With Hypophosphatasia Treated With Asfotase Alfa. Cornea. 2019 Jul;38(7):896-900. doi: 10.1097/ICO.0000000000001947. PMID 30969260
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Healthcare Providers — http://www.hypophosphatasia.com/hcp/

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.3 mg/kg Asfotase Alfa: Asfotase alfa Cohort 1: Daily SC injections of 0.3 mg/kg asfotase alfa (2.1 mg/kg/week total).
  Following completion of the Week 24 visit, all subjects were eligible to participate in an open-label extension treatment period. In this extension period, all subjects were treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects received 1 mg/kg/day 6 days/week until regulatory approval of the drug.
- 0.5 mg/kg Asfotase Alfa: Asfotase alfa Cohort 2: Daily SC injections of 0.5 mg/kg asfotase alfa (3.5 mg/kg/week total).
  Following completion of the Week 24 visit, all subjects were eligible to participate in an open-label extension treatment period. In this extension period, all subjects were treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects received 1 mg/kg/day 6 days/week until regulatory approval of the drug.
- Concurrent Control: No asfotase alfa during first 24 weeks (primary treatment period).
  Following completion of the Week 24 visit, all subjects were eligible to participate in an open-label extension treatment period. In this extension period, all subjects were treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects received 1 mg/kg/day 6 days/week until regulatory approval of the drug.
Period: Primary Treatment Period
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control
Started | 7 | 6 | 6
Completed | 7 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Extension Treatment Period
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control
Started | 7 | 6 | 6
Completed | 5 | 5 | 4
Not Completed | 2 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Noncompliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All efficacy analyses were performed on the full analysis set (intent-to-treat population), which consisted of all randomized patients (n=19).
Groups:
- 0.3 mg/kg Asfotase Alfa: Asfotase alfa: Cohort 1: Daily SC injections of 0.3 mg/kg asfotase alfa (total of 2.1 mg/kg/week) during Primary Treatment Period through Week 24.
  Following completion of the Week 24 visit, all subjects were eligible to participate in an open-label extension treatment period. In this extension period, all subjects were treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects received 1 mg/kg/day 6 days/week until regulatory approval of the drug.
- 0.5 mg/kg Asfotase Alfa: Asfotase alfa: Cohort 2: Daily SC injections of 0.5 mg/kg asfotase alfa (3.5 mg/kg/week total) during Primary Treatment Period through Week 24.
  Following completion of the Week 24 visit, all subjects were eligible to participate in an open-label extension treatment period. In this extension period, all subjects were treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects received 1 mg/kg/day 6 days/week until regulatory approval of the drug.
- Concurrent Control: No asfotase alfa during first 24 weeks (primary treatment period).
  Following completion of the Week 24 visit, all subjects randomized to the concurrent control cohort were eligible to participate in an open-label extension treatment period. In this extension period, all subjects were treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects received 1 mg/kg/day 6 days/week until regulatory approval of the drug
- Total: Total of all reporting groups
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Total
Number analyzed (Participants) | 7 | 6 | 6 | 19
Age, Continuous [Median (Full Range); unit: years] | 45.0 [14 to 66] | 55.0 [15 to 57] | 21.0 [13 to 58] | 53.0 [13 to 66]
Age, Customized [Median (Full Range); unit: years]
  Age at Onset of Symptoms | 2.0 [0.2 to 36] | 2.0 [0 to 3] | 0.88 [0.2 to 4.0] | 2.0 [0 to 36]
Age, Customized [Count of Participants; unit: Participants]
  Age Group: Adolescent (12-17 years) | 2 | 1 | 3 | 6
  Age Group: Adult (≥ 18 years) | 5 | 5 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 12
  Male | 1 | 2 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 6 | 5 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Hypophosphatasia (HPP) Phenotype [Count of Participants; unit: Participants]
  Infantile (<6 months) | 1 | 2 | 1 | 4
  Juvenile (≥ 6 months to < 18 years) | 5 | 4 | 5 | 14
  Adult (≥ 18 years) | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 for Plasma Pyridoxal-5' Phosphate (PLP)
Description: Blood samples were collected to evaluate the effect of asfotase alfa on reduction in plasma pyridoxal-5' phosphate (PLP)
Time Frame: Baseline, Week 24
Population: Full analysis set (intent-to-treat, all randomized patients)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 0.3 mg/kg Asfotase Alfa: Asfotase alfa Cohort 1: Daily SC injections of 0.3 mg/kg asfotase alfa (2.1 mg/kg/week total)
- 0.5 mg/kg Asfotase Alfa: Asfotase alfa Cohort 2: Daily SC injections of 0.5 mg/kg asfotase alfa (3.5 mg/kg/week total)
- Concurrent Control: Control (no asfotase alfa) during primary treatment period (first 24 weeks)
- Combined Asfotase Alfa Group: Subjects from Cohort 1 and Cohort 2 treated with asfotase alfa during primary treatment period (first 24 weeks)
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Combined Asfotase Alfa Group
Number analyzed (Participants) | 7 | 6 | 6 | 13
ng/mL | -254.96 (196.206) | -564.27 (624.009) | 3.13 (242.721) | -397.72 (455.249)
Statistical Analysis 1: Comparison: Concurrent Control vs Combined Asfotase Alfa Group; PLP Change from Baseline to Week 24; Test type: Superiority — If p-values were less than 0.05 and the Hodges-Lehman-Sen estimate favored asfotase alfa (eg, it had a negative sign indicating the between-group differences in change from Baseline favored treated patients), then superiority over control was claimed; p = 0.0285, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehman-Sen = -302.05, 95% CI 2-sided [-626.40 to -59.20]

2. Primary Outcome: Change From Baseline to Week 24 for Plasma Inorganic Pyrophosphate (PPi)
Description: Blood samples were collected to evaluate the effect of asfotase alfa on reduction in plasma inorganic pyrophosphate (PPi)
Time Frame: Baseline, Week 24
Population: Full analysis set (intent-to-treat, all randomized patients)
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Combined Asfotase Alfa Group
Number analyzed (Participants) | 7 | 6 | 6 | 13
uM | -2.027 (1.4381) | -2.185 (1.3304) | -1.052 (2.9248) | -2.100 (1.3335)
Statistical Analysis 1: Comparison: Concurrent Control vs Combined Asfotase Alfa Group; PPi Change from Baseline to Week 24; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0715, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehman-Sen = -1.825, 95% CI 2-sided [-3.210 to 0.230] — Estimate and exact confidence interval are from Hodges-Lehmann-Sen method for location shift in distribution between the treatment group and the control group

3. Primary Outcome: Safety and Tolerability of Asfotase Alfa
Description: The safety and tolerability of daily subcutaneous (SC) injections of asfotase alfa was assessed by routine monitoring of patients for treatment-emergent adverse events (TEAEs) and injection-associated reactions (IARs).
Time Frame: Up to 288 weeks exposure to asfotase alfa
Population: Safety Set. Control group and asfotase alfa Cohorts during the primary treatment period (first 24 weeks of study); all patients with asfotase alfa exposure during open-label extension treatment period.
Measure: Number; unit: Number of Treatment-Emergent Events
Groups:
- 0.3 mg/kg Asfotase Alfa: Primary Treatment Period (first 24 week). Asfotase alfa Cohort 1: Daily SC injections of 0.3 mg/kg asfotase alfa (2.1 mg/kg/week total).
- 0.5 mg/kg Asfotase Alfa: Primary Treatment Period (first 24 weeks). Asfotase alfa Cohort 2: Daily SC injections of 0.5 mg/kg asfotase alfa (3.5 mg/kg/week total).
- Concurrent Control: No asfotase alfa during primary treatment period: (first 24 weeks).
- Cumulative Exposure to Asfotase Alfa: All subjects from Cohort 1, Cohort 2, or Control group with any asfotase alfa exposure. During primary treatment period, N=13. During open-label extension treatment period, N=19.
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Cumulative Exposure to Asfotase Alfa
Number analyzed (Participants) | 7 | 6 | 6 | 19
Number of Treatment-Emergent Events
  Any TEAE | 243 | 81 | 45 | 1145
  Not related TEAEs | 110 | 69 | 45 | 731
  Related TEAEs | 133 | 12 | 0 | 414
  Injection site reactions | 133 | 12 | 0 | 385
  Serious TEAEs | 1 | 1 | 4 | 29
  TEAEs leading to withdrawal | 0 | 0 | 0 | 2
  Deaths | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Bone Mineral Content (BMC) as Measured by Dual-energy X-ray Absorptiometry (DXA)
Description: A DXA scan was performed to evaluate bone mineral content (BMC) of the spine, hip, and whole body during the primary (first 24 weeks) and extension treatment periods (up to 288 weeks).
Time Frame: Baseline, every 24 weeks through Week 96, then every 48 weeks until Week 288.
Population: Full analysis set (intent-to-treat, all randomized patients)
Measure: Mean (Standard Deviation); unit: g
Groups:
- Asfotase Alfa Combined: All subjects from Cohort 1, Cohort 2, or Control group with any asfotase alfa exposure. During primary treatment period, N=13. During open-label extension treatment period, N=19.
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Asfotase Alfa Combined
Number analyzed (Participants) | 7 | 6 | 6 | 19
g
  Hip total BMC Week 24: number analyzed (Participants) | 4 | 5 | 4 | 9
  Hip total BMC Week 24 | -3.288 (7.7669) | 1.214 (2.2154) | 1.288 (0.9161) | -0.787 (5.5411)
  Hip total BMC Week 48: number analyzed (Participants) | 1 | 1 | 4 | 6
  Hip total BMC Week 48 | 1.160 (NA) — Data available for only 1 subject | 4.530 (NA) — Data available for only 1 subject | 2.320 (1.3990) | 2.495 (1.5438)
  Hip total BMC Week 96: number analyzed (Participants) | 4 | 4 | 3 | 11
  Hip total BMC Week 96 | 0.082 (1.4046) | 4.345 (4.0466) | 2.907 (2.0087) | 2.403 (3.1702)
  Hip total BMC Week 144: number analyzed (Participants) | 3 | 4 | 3 | 10
  Hip total BMC Week 144 | 1.630 (1.8719) | 5.043 (5.5955) | 4.533 (1.4621) | 3.866 (3.7577)
  Hip total BMC Week 192: number analyzed (Participants) | 2 | 4 | 3 | 9
  Hip total BMC Week 192 | 1.080 (2.0082) | 4.725 (6.4843) | 2.910 (0.2910) | 3.310 (4.3124)
  Hip total BMC Week 240: number analyzed (Participants) | 2 | 3 | 3 | 8
  Hip total BMC Week 240 | 0.550 (2.4042) | 6.807 (5.7557) | -0.673 (0.1644) | 2.438 (4.8626)
  Hip Total BMC Week 288: number analyzed (Participants) | 0 | 1 | 0 | 1
  Hip Total BMC Week 288 |  | -2.780 (NA) — Data available for only 1 subject |  | -2.780 (NA) — Data available for only 1 subject
  Hip Total BMC Last Overall Exposure: number analyzed (Participants) | 4 | 5 | 4 | 13
  Hip Total BMC Last Overall Exposure | 0.080 (1.8713) | 3.604 (5.8284) | 0.328 (2.0062) | 1.512 (4.0224)
  Lumbar Spine BMC Week 24: number analyzed (Participants) | 7 | 5 | 5 | 12
  Lumbar Spine BMC Week 24 | 2.477 (2.5616) | 2.768 (2.0007) | 1.432 (1.7824) | 2.598 (2.2488)
  Lumbar Spine BMC Week 48: number analyzed (Participants) | 1 | 1 | 5 | 7
  Lumbar Spine BMC Week 48 | 2.420 (NA) — Data available for only 1 subject | 5.550 (NA) — Data available for only 1 subject | 4.842 (5.7882) | 4.597 (4.8298)
  Lumbar Spine BMC Week 96: number analyzed (Participants) | 7 | 5 | 4 | 16
  Lumbar Spine BMC Week 96 | 3.356 (4.4566) | 4.174 (3.7068) | 7.330 (5.6953) | 4.605 (4.5680)
  Lumbar Spine BMC Week 144: number analyzed (Participants) | 5 | 5 | 4 | 14
  Lumbar Spine BMC Week 144 | 2.086 (5.2198) | 5.828 (3.9791) | 6.710 (4.0174) | 4.744 (4.6193)
  Lumbar Spine BMC Week 192: number analyzed (Participants) | 5 | 5 | 4 | 14
  Lumbar Spine BMC Week 192 | 2.094 (16.4419) | 6.162 (4.1628) | 5.197 (5.7568) | 4.434 (9.9797)
  Lumbar Spine BMC Week 240: number analyzed (Participants) | 5 | 4 | 4 | 13
  Lumbar Spine BMC Week 240 | 3.536 (17.0957) | 3.298 (2.4931) | 5.037 (4.7161) | 3.925 (10.2539)
  Lumbar Spine BMC Week 288: number analyzed (Participants) | 1 | 1 | 0 | 2
  Lumbar Spine BMC Week 288 | 20.190 (NA) — Data available for only 1 subject | 6.500 (NA) — Data available for only 1 subject |  | 13.705 (10.1894)
  Lumbar Spine BMC Last Overall Exposure: number analyzed (Participants) | 7 | 5 | 5 | 17
  Lumbar Spine BMC Last Overall Exposure | 4.306 (14.5714) | 5.130 (3.5930) | 6.714 (5.1113) | 5.256 (9.5103)
  Whole Body BMC Week 24: number analyzed (Participants) | 7 | 5 | 5 | 12
  Whole Body BMC Week 24 | -21.871 (35.4370) | 41.454 (20.0358) | 237.248 (414.0877) | 4.514 (43.5228)
  Whole Body BMC Week 48: number analyzed (Participants) | 1 | 1 | 5 | 7
  Whole Body BMC Week 48 | 49.820 (NA) — Data available for only 1 subject | 72.530 (NA) — Data available for only 1 subject | 30.228 (82.4369) | 39.070 (69.2934)
  Whole Body BMC Week 96: number analyzed (Participants) | 7 | 5 | 4 | 16
  Whole Body BMC Week 96 | 7.537 (74.2838) | 59.604 (97.9214) | 98.018 (111.9259) | 46.428 (93.5046)
  Whole Body BMC Week 144: number analyzed (Participants) | 5 | 5 | 4 | 14
  Whole Body BMC Week 144 | -48.236 (111.6604) | 17.446 (173.3574) | 92.063 (107.9837) | 15.307 (138.3534)
  Whole Body BMC Week 192: number analyzed (Participants) | 5 | 5 | 4 | 14
  Whole Body BMC Week 192 | -121.916 (92.0001) | 23.938 (195.8402) | 50.375 (99.6281) | -20.599 (151.5153)
  Whole Body BMC Week 240: number analyzed (Participants) | 5 | 4 | 4 | 13
  Whole Body BMC Week 240 | -97.706 (106.6581) | 82.310 (223.0794) | 40.572 (162.1575) | 0.231 (172.0218)
  Whole Body BMC Week 288: number analyzed (Participants) | 1 | 1 | 0 | 2
  Whole Body BMC Week 288 | -243.080 (NA) — Data available for only 1 subject | -144.660 (NA) — Data available for only 1 subject |  | -193.870 (69.5934)
  Whole Body BMC Last Overall Exposure: number analyzed (Participants) | 7 | 5 | 5 | 17
  Whole Body BMC Last Overall Exposure | -113.296 (178.8050) | 11.252 (217.5674) | 82.548 (128.7017) | -19.063 (188.0498)
Statistical Analysis 1: Comparison: Concurrent Control vs Asfotase Alfa Combined; Hip Total BMC Change from Baseline to Week 24; Test type: Superiority; p = 0.3301, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehmann-Sen = -0.910, 95% CI 2-sided [-3.320 to 1.780]
Statistical Analysis 2: Comparison: Concurrent Control vs Asfotase Alfa Combined; Lumbar Spine BMC Change from Baseline to Week 24; Test type: Superiority; p = 0.3827, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehmann-Sen = 1.330, 95% CI 2-sided [-1.360 to 3.120]
Statistical Analysis 3: Comparison: Concurrent Control vs Asfotase Alfa Combined; Whole Body BMC Change from Baseline to Week 24; Test type: Superiority; p = 0.0485, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehmann-Sen = -77.100, 95% CI 2-sided [-917.440 to -1.740]

5. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) as Measured by Dual-energy X-ray Absorptiometry (DXA)
Description: A DXA scan was performed to evaluate bone bone mineral density (BMD) of the spine, hip, and whole body during the primary (first 24 weeks) and extension treatment periods (up to 288 weeks).
Time Frame: Baseline, every 24 weeks through Week 96, then every 48 weeks until Week 288.
Population: Full analysis set (intent-to-treat, all randomized patients)
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Asfotase Alfa Combined
Number analyzed (Participants) | 7 | 6 | 6 | 19
g/cm2
  Hip total BMD Week 24: number analyzed (Participants) | 4 | 5 | 4 | 9
  Hip total BMD Week 24 | 0.0477 (0.07710) | 0.0094 (0.02441) | 0.0195 (0.01642) | 0.0251 (0.05361)
  Hip total BMD Week 48: number analyzed (Participants) | 1 | 1 | 4 | 6
  Hip total BMD Week 48 | 0.0190 (NA) — Data available for only 1 subject | 0.0240 (NA) — Data available for only 1 subject | 0.0590 (0.04109) | 0.0465 (0.03729)
  Hip total BMD Week 96: number analyzed (Participants) | 4 | 4 | 3 | 11
  Hip total BMD Week 96 | 0.0003 (0.00532) | 0.0780 (0.06703) | 0.0480 (0.04943) | 0.0415 (0.05542)
  Hip total BMD Week 144: number analyzed (Participants) | 3 | 4 | 3 | 10
  Hip total BMD Week 144 | 0.0340 (0.02524) | 0.0923 (0.07682) | 0.0933 (0.04150) | 0.0751 (0.05741)
  Hip total BMD Week 192: number analyzed (Participants) | 2 | 4 | 3 | 9
  Hip total BMD Week 192 | 0.0135 (0.00919) | 0.0983 (0.10856) | 0.0563 (0.07100) | 0.0654 (0.08327)
  Hip total BMD Week 240: number analyzed (Participants) | 2 | 3 | 3 | 8
  Hip total BMD Week 240 | 0.0115 (0.02192) | 0.1137 (0.05701) | -0.0073 (0.06178) | 0.0428 (0.07481)
  Hip total BMD Week 288: number analyzed (Participants) | 0 | 1 | 0 | 1
  Hip total BMD Week 288 |  | -0.0200 (NA) — Data available for only 1 subject |  | -0.0200 (NA) — Data available for only 1 subject
  Hip total BMD Last Overall Exposure: number analyzed (Participants) | 4 | 5 | 4 | 13
  Hip total BMD Last Overall Exposure | -0.0115 (0.03899) | 0.0658 (0.07776) | 0.0207 (0.07549) | 0.0282 (0.07038)
  Lumbar Spine BMD Week 24: number analyzed (Participants) | 7 | 5 | 5 | 12
  Lumbar Spine BMD Week 24 | 0.0269 (0.02113) | 0.0272 (0.01492) | 0.0098 (0.02475) | 0.0270 (0.01802)
  Lumbar Spine BMD Week 48: number analyzed (Participants) | 1 | 1 | 5 | 7
  Lumbar Spine BMD Week 48 | 0.0480 (NA) — Data available for only 1 subject | 0.0590 (NA) — Data available for only 1 subject | 0.0914 (0.05647) | 0.0806 (0.04978)
  Lumbar Spine BMD Week 96: number analyzed (Participants) | 7 | 5 | 4 | 16
  Lumbar Spine BMD Week 96 | 0.0414 (0.05230) | 0.0554 (0.04271) | 0.1158 (0.08060) | 0.0644 (0.06210)
  Lumbar Spine BMD Week 144: number analyzed (Participants) | 5 | 5 | 4 | 14
  Lumbar Spine BMD Week 144 | 0.0200 (0.06257) | 0.0850 (0.05323) | 0.1138 (0.05734) | 0.0700 (0.06688)
  Lumbar Spine BMD Week 192: number analyzed (Participants) | 5 | 5 | 4 | 14
  Lumbar Spine BMD Week 192 | 0.0554 (0.13220) | 0.0766 (0.04180) | 0.1123 (0.05197) | 0.0792 (0.08423)
  Lumbar Spine BMD Week 240: number analyzed (Participants) | 5 | 4 | 4 | 13
  Lumbar Spine BMD Week 240 | 0.0750 (0.14168) | 0.0455 (0.04107) | 0.1027 (0.04786) | 0.0745 (0.09073)
  Lumbar Spine BMD Week 288: number analyzed (Participants) | 1 | 1 | 0 | 2
  Lumbar Spine BMD Week 288 | 0.1860 (NA) — Data available for only 1 subject | 0.0700 (NA) — Data available for only 1 subject |  | 0.1280 (0.08202)
  Lumbar Spine BMD Last Overall Exposure: number analyzed (Participants) | 7 | 5 | 5 | 17
  Lumbar Spine BMD Last Overall Exposure | 0.0737 (0.11346) | 0.0492 (0.04649) | 0.1194 (0.04999) | 0.0799 (0.08241)
  Whole Body BMD Week 24: number analyzed (Participants) | 7 | 5 | 5 | 12
  Whole Body BMD Week 24 | -0.0003 (0.01788) | -0.0122 (0.01055) | 0.0206 (0.03173) | -0.0052 (0.01589)
  Whole Body BMD Week 48: number analyzed (Participants) | 1 | 1 | 5 | 7
  Whole Body BMD Week 48 | 0.0050 (NA) — Data available for only 1 subject | 0.0090 (NA) — Data available for only 1 subject | 0.0178 (0.05277) | 0.0147 (0.04342)
  Whole Body BMD Week 96: number analyzed (Participants) | 7 | 5 | 4 | 16
  Whole Body BMD Week 96 | -0.0103 (0.03523) | -0.0100 (0.04136) | 0.0230 (0.04872) | -0.0019 (0.04059)
  Whole Body BMD Week 144: number analyzed (Participants) | 5 | 5 | 4 | 14
  Whole Body BMD Week 144 | -0.0250 (0.03662) | -0.0278 (0.05823) | -0.0060 (0.04721) | -0.0206 (0.04542)
  Whole Body BMD Week 192: number analyzed (Participants) | 5 | 5 | 4 | 14
  Whole Body BMD Week 192 | -0.0532 (0.02477) | -0.0220 (0.07088) | -0.0212 (0.06209) | -0.0329 (0.05358)
  Whole Body BMD Week 240: number analyzed (Participants) | 5 | 4 | 4 | 13
  Whole Body BMD Week 240 | -0.0426 (0.05601) | -0.0122 (0.08610) | -0.0493 (0.06965) | -0.0353 (0.06615)
  Whole Body BMD Week 288: number analyzed (Participants) | 1 | 1 | 0 | 2
  Whole Body BMD Week 288 | -0.1140 (NA) — Data available for only 1 subject | -0.0710 (NA) — Data available for only 1 subject |  | -0.0925 (0.03041)
  Whole Body BMD Last Overall Exposure: number analyzed (Participants) | 7 | 5 | 5 | 17
  Whole Body BMD Last Overall Exposure | -0.0501 (0.07360) | -0.0298 (0.08785) | -0.0224 (0.05773) | -0.0360 (0.07036)
Statistical Analysis 1: Comparison: Concurrent Control vs Asfotase Alfa Combined; Hip Total Change from Baseline to Week 24; Test type: Superiority; p = 0.7357, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehmann-Sen = -0.0125, 95% CI 2-sided [-0.0400 to 0.0390]
Statistical Analysis 2: Comparison: Concurrent Control vs Asfotase Alfa Combined; Lumbar Spine BMD Change from Baseline to Week 24; Test type: Superiority; p = 0.2439, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehmann-Sen = 0.0255, 95% CI 2-sided [-0.0090 to 0.0410]
Statistical Analysis 3: Comparison: Concurrent Control vs Asfotase Alfa Combined; Whole Body BMD Change from Baseline to Week 24; Test type: Superiority; p = 0.1222, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehmann-Sen = -0.0315, 95% CI 2-sided [-0.0590 to 0.0120]

6. Secondary Outcome: Change in Walking Ability as Measured by the Six-Minute Walk Test (6MWT)
Description: The patient was instructed to walk the length of a pre-measured hallway for 6 minutes. The primary measurement was distance walked (in meters).
Time Frame: Baseline, Week 24 (primary treatment period) and up to 288 weeks of asfotase alfa exposure
Population: Full analysis set (intent-to-treat, all randomized patients). Among the 6 control subjects, only 4 had both a Baseline and Week 24 value.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- 0.3 mg/kg Asfotase Alfa: Asfotase alfa Cohort 1: Daily SC injections of 0.3 mg/kg asfotase alfa (2.1 mg/kg/week total) during Primary Treatment Period through Week 24.
  Following completion of the Week 24 visit, all subjects were eligible to participate in an open-label extension treatment period. In this extension period, all subjects were treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects received 1 mg/kg/day 6 days/week until regulatory approval of the drug.
- 0.5 mg/kg Asfotase Alfa: Asfotase alfa Cohort 2: Daily SC injections of 0.5 mg/kg asfotase alfa (3.5 mg/kg/week total) during Primary Treatment Period through Week 24.
  Following completion of the Week 24 visit, all subjects were eligible to participate in an open-label extension treatment period. In this extension period, all subjects were treated with daily SC injections of 0.5 mg/kg/day asfotase alfa (a total of 3.5 mg/kg/week) for approximately 24 weeks, then subjects received 1 mg/kg/day 6 days/week until regulatory approval of the drug.
- Asfotase Alfa Combined: Subjects From Cohort 1 and Cohort 2 treated with asfotase alfa (N=13) during Primary Treatment Period, and all subjects exposed to asfotase alfa (N=19) during extension treatment period.
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Asfotase Alfa Combined
Number analyzed (Participants) | 7 | 6 | 6 | 19
meters
  Change from Baseline to Week 24: number analyzed (Participants) | 7 | 6 | 4 | 13
  Change from Baseline to Week 24 | 64.7 (73.04) | 43.5 (43.18) | 13.5 (69.77) | 54.9 (59.71)
  Change from Baseline Last Overall Exposure: number analyzed (Participants) | 7 | 6 | 5 | 18
  Change from Baseline Last Overall Exposure | 89.4 (81.32) | 2.2 (121.79) | 74.4 (107.40) | 56.2 (104.85)
Statistical Analysis 1: Comparison: Concurrent Control vs Asfotase Alfa Combined; Week 24 Change from Baseline; Test type: Superiority; p = 0.1303, Wilcoxon rank-sum — Two-sided with p-value threshold <0.05 for statistical significance; Hodges-Lehmann-Sen = 44.0, 95% CI 2-sided [-73.0 to 114.0] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change From Baseline in HPP-related Osteomalacia as Measured by Trans-iliac Crest Bone Biopsy: Osteoid Volume/Bone Volume
Description: A trans-iliac crest bone biopsy was performed to quantify changes from Baseline in histomorphometric parameters relevant for evaluation of osteomalacia severity, including Osteoid Volume/Bone Volume (%). The difference in time under observation between asfotase alfa groups (Week 48) and control group (Week 24) resulted from study design, ie, control subjects transitioned to active treatment after the Week 24 visit.
Time Frame: Baseline, Week 24 (Control group), and Week 48 (Asfotase alfa groups).
Population: Full analysis set (intent-to-treat, all randomized patients)
Measure: Mean (Standard Deviation); unit: percentage of volume
Groups:
- Asfotase Alfa Combined: Subjects from primary treatment period asfotase alfa groups.
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Asfotase Alfa Combined
Number analyzed (Participants) | 6 | 6 | 6 | 12
percentage of volume | 1.213 (3.2488) | -2.845 (2.3769) | 0.200 (4.7679) | -0.816 (3.4434)

8. Secondary Outcome: Change From Baseline in HPP-related Osteomalacia as Measured by Trans-iliac Crest Bone Biopsy: Osteoid Thickness
Description: A trans-iliac crest bone biopsy was performed to quantify changes from Baseline in histomorphometric parameters relevant for evaluation of osteomalacia severity, including Osteoid Thickness (um). The difference in time under observation between asfotase alfa groups (Week 48) and control group (Week 24) resulted from study design, ie, control subjects transitioned to active treatment after the Week 24 visit.
Time Frame: Baseline, Week 24 (Control group), and Week 48 (Asfotase alfa groups).
Population: Full analysis set (intent-to-treat, all randomized patients)
Measure: Mean (Standard Deviation); unit: um
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Asfotase Alfa Combined
Number analyzed (Participants) | 6 | 6 | 6 | 12
um | -0.013 (3.6333) | -1.516 (2.3556) | -1.132 (6.0884) | -0.764 (3.0229)

9. Secondary Outcome: Change From Baseline in HPP-related Osteomalacia as Measured by Trans-iliac Crest Bone Biopsy: Mineralization Lag Time
Description: A trans-iliac crest bone biopsy was performed to quantify changes from Baseline in histomorphometric parameters relevant for evaluation of osteomalacia severity, including Mineralization Lag Time (days). The difference in time under observation between asfotase alfa groups (Week 48) and control group (Week 24) resulted from study design, ie, control subjects transitioned to active treatment after the Week 24 visit.
Time Frame: Baseline, Week 24 (Control group), and Week 48 (Asfotase alfa groups).
Population: Full analysis set (intent-to-treat, all randomized patients)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 0.3 mg/kg Asfotase Alfa | 0.5 mg/kg Asfotase Alfa | Concurrent Control | Asfotase Alfa Combined
Number analyzed (Participants) | 4 | 5 | 5 | 9
days | -908.255 (1313.6158) | -126.946 (142.2929) | 78.296 (167.0895) | -474.195 (909.2779)

ADVERSE EVENTS:
Time Frame: up to 288 weeks
Description: Only adverse events with an onset date are included in the cumulative exposure category.
Groups:
- 0.3 mg/kg Asfotase Alfa (First 24 Weeks): Asfotase alfa Cohort 1: Daily SC injections of 0.3 mg/kg asfotase alfa (2.1 mg/kg/week total)
- 0.5 mg/kg Asfotase Alfa (First 24 Weeks): Asfotase alfa Cohort 2: Daily SC injections of 0.5 mg/kg asfotase alfa (3.5 mg/kg/week total)
- Concurrent Control (First 24 Weeks): No asfotase alfa treatment during primary treatment period: first 24 weeks.
  After 24 weeks, Control Group subjects were eligible to begin asfotase alfa treatment in the open-label extension treatment period.
- Cumulative Exposure to Asfotase Alfa: Adverse events occurring in subjects from Cohort 1, Cohort 2 and original Control group during exposure to asfotase alfa.
Arm/Group | 0.3 mg/kg Asfotase Alfa (First 24 Weeks) | 0.5 mg/kg Asfotase Alfa (First 24 Weeks) | Concurrent Control (First 24 Weeks) | Cumulative Exposure to Asfotase Alfa
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/6 | 2/6 | 9/19
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 6/6 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg/kg Asfotase Alfa (First 24 Weeks) (N=7) | 0.5 mg/kg Asfotase Alfa (First 24 Weeks) (N=6) | Concurrent Control (First 24 Weeks) (N=6) | Cumulative Exposure to Asfotase Alfa (N=19)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial Pressure Increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Device Dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arnold-Chiari Malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactoid Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg/kg Asfotase Alfa (First 24 Weeks) (N=7) | 0.5 mg/kg Asfotase Alfa (First 24 Weeks) (N=6) | Concurrent Control (First 24 Weeks) (N=6) | Cumulative Exposure to Asfotase Alfa (N=19)
Injection Site Erythema (General disorders) | 3 (61) | 2 (5) | 0 (0) | 13 (121)
Injection Site Haematoma (General disorders) | 3 (14) | 1 (6) | 0 (0) | 10 (33)
Injection Site Pain (General disorders) | 4 (20) | 0 (0) | 0 (0) | 6 (26)
Fatigue (General disorders) | 0 (0) | 3 (5) | 0 (0) | 4 (7)
Injection Site Pruritis (General disorders) | 3 (16) | 0 (0) | 0 (0) | 5 (20)
Injection Site Discoloration (General disorders) | 2 (9) | 0 (0) | 0 (0) | 9 (66)
Injection Site Swelling (General disorders) | 2 (10) | 0 (0) | 0 (0) | 4 (12)
Oedema Peripheral (General disorders) | 1 (7) | 1 (1) | 0 (0) | 8 (16)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Facial Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Feeling Abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection Site Induration (General disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (4)
Injection Site Papule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Local Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Medical Device Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection Site Atrophy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Injection Site Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (56)
Injection Site Warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 1 (3) | 10 (14)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 (7) | 3 (3) | 0 (0) | 7 (16)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (13) | 3 (7) | 1 (1) | 12 (46)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 2 (3) | 1 (2) | 13 (41)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2) | 0 (0) | 9 (14)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (4) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 8 (11)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (3) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Nodule On Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 2 (5)
Deformity Thorax (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tendon Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 6 (8)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 5 (20)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 7 (22)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinea Pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (5)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 1 (1) | 5 (28)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (7)
Dizziness Exertional (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (5)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (9)
Post-Traumatic Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 5 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (2) | 4 (7)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tooth Loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Blood human Chorionic Gonadotropin Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood Parathyroid Hormone Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Heart Rate Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Vitamin D Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (8)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (8) | 0 (0) | 0 (0) | 1 (8)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash Macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 5 (8)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 7 (10)
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Post Procedural Swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (3) | 5 (11)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear Discomfort (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Ear Pruritis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lacrimation Increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Deposit (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Keratopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food Allergy (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Gout (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (7)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection Site Hypertrophy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (12)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Loose Tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Deposit Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Vitreous Detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Optic Atrophy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Initial Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breast Calcifications (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breast Mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Axillary Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Catherter Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Catheter SIte Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (17)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device Failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection Site Exfoliation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Macule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (10)
Injection Site Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection Site Scar (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Joint Warmth (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower Extremity Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ilium Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Procedural Nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal Mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic Polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival Hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Adenovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Conjunctivitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Staphylococcal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tinea Cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning Sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial Pressure Increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excessive Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrown Hair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Conjunctival Discolouration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival Disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal Deposits (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid Disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Punctate Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial Hypereactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood 25-Hydroxycholecalciferol Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Alkaline Phoshatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemaglobin Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart Rate Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Physical Examination Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red Blood Cells Urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ultrasound Kidney Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional Self-Injury (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spermatocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen Impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tympanic Membrane Disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon Polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunisation Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less